CLINICAL TRIAL: NCT06952712
Title: Aspirin 150 mg vs 100 mg for Prevention of Preeclampsia in High-Risk Obese Pregnant Women: A Multicenter Randomized Controlled Trial
Brief Title: Aspirin 150 mg vs 100 mg for Prevention of Preeclampsia in High-Risk Obese Pregnant Women
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: FANG HE (Other)
Responsible Party: Sponsor-Investigator, FANG HE, Chief Physician/Professor of the Obstetrics Department, The Third Affiliated Hospital of Guangzhou Medical University
Organization: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: [2025] Ethics Review NO.059
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Preeclampsia
Keywords: Low-dose aspirin; preeclampsia; obese; pregnant women; randomized controlled trial
MeSH Terms: conditions — Pre-Eclampsia; Obesity | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Obese pregnant women with normal NT scan results and risk factors for preeclampsia were included. They were randomly assigned in a 1:1 ratio at 12-16 weeks of gestation. The control group took 100 mg of aspirin orally every night, while the experimental group took 150 mg of aspirin orally every night, until 36+0 to 36+6 weeks of gestation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin 100mg (Active Comparator): Aspirin 100mg qn was started from 12-16 weeks of gestation and discontinued from 36+0-36+6 weeks of gestation
  Interventions: Drug: Aspirin 100mg
- Aspirin 150mg (Experimental): Aspirin 150mg qn was started from 12-16 weeks of gestation and discontinued from 36+0-36+6 weeks of gestation
  Interventions: Drug: Aspirin 150mg

INTERVENTIONS:
Drug: Aspirin 100mg — Aspirin 100mg qn was started from 12-16 weeks of gestation and discontinued from 36+0-36+6 weeks of gestation
  Arms: Aspirin 100mg
Drug: Aspirin 150mg — Aspirin 150mg qn was started from 12-16 weeks of gestation and discontinued from 36+0-36+6 weeks of gestation
  Arms: Aspirin 150mg

SUMMARY:
According to the American College of Obstetricians and Gynecologists (ACOG), pregnancy-induced hypertension is defined as a new onset of systolic and/or diastolic blood pressure ≥140/90 mmHg after 20 weeks of gestation, with at least 4 hours between two blood pressure measurements, and blood pressure can return to normal after childbirth. Preeclampsia is defined as the presence of proteinuria or multi-organ dysfunction on the basis of pregnancy-induced hypertension. Obese women are a high-risk group for preeclampsia, and the preventive use of low-dose aspirin (LDA) is one of the currently recognized effective interventions. Obesity, as an independent risk factor for preeclampsia, can increase the risk of the disease by 2 to 3 times. With the rising global obesity rate, the prevention and control of preeclampsia in obese pregnant women has become an important challenge in the field of perinatal medicine. The WHO report indicates that the incidence of preeclampsia in obese women is significantly higher, with a 20-30% increase in preeclampsia risk for every 5-unit increase in BMI. The incidence of preeclampsia in obese women can reach 15-25%. At present, the clinical application of oral aspirin for the prevention of preeclampsia in China mainly follows authoritative consensuses such as the "Guidelines for the Diagnosis and Treatment of Hypertensive Disorders in Pregnancy (2020)", which recommends that high-risk pregnant women (such as those with obesity, chronic hypertension, and a history of preeclampsia in the previous pregnancy) take low-dose aspirin (50-150 mg/d) orally from 12 to 16 weeks of gestation for prevention. However, in actual clinical practice, a dose of 100 mg/d is commonly used, and there is still a lack of clear guidance on whether the dose needs to be adjusted for obese pregnant women. At present, the dose of aspirin mainly used in China is still 100 mg, while foreign studies are more inclined to use 150 mg. Therefore, this study is designed to conduct a randomized controlled trial to compare the efficacy and safety of 100 mg and 150 mg aspirin in preventing preeclampsia in obese pregnant women, to optimize the LDA strategy for the prevention of preeclampsia and provide high-quality evidence for clinical practice.

DETAILED DESCRIPTION:
This study aims to compare the efficacy and safety of 100 mg and 150 mg aspirin in preventing preeclampsia in obese pregnant women and to optimize the LDA strategy for the prevention of preeclampsia. Obese pregnant women at high risk of preeclampsia will be randomly assigned in a 1:1 ratio at 12-16 weeks of gestation. The control group will take 100 mg of aspirin orally every night, while the experimental group will take 150 mg of aspirin orally every night, until 36+0 to 36+6 weeks of gestation. The incidence of preeclampsia will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years;
2. Pregnancy 12-16 weeks, NT normal;
3. Singleton pregnancy;
4. a.BMI ≥35kg/m²; b. 28≤BMI <35 kg/m², and at least one risk factor: history of preeclampsia, chronic hypertension, type 1 or type 2 diabetes, autoimmune disease (excluding antiphospholipid syndrome), nulliparous, family history of preeclampsia, placental abruption, stillbirth, SGA, more than 10 years between pregnancies, in vitro fertilization-embryo transfer;
5. Sign informed consent

Exclusion Criteria:

* 1. Aspirin allergy or contraindication (such as active gastric ulcer, coagulation disorder); 2. Multiple pregnancies; 3. Other severe comorbidities that may lead to pregnancy complications; 4. Seizures; 5. Renal disease, baseline proteinuria (proteinuria> 3+, or protein-to-creatinine ratio ≥ 0.3); 6. Patients taking aspirin for other reasons (such as stroke, heart disease)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1300 (Estimated)
Dates: Start 2025-05-07 (Estimated); Primary Completion 2028-05-06 (Estimated); Study Completion 2028-05-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of preeclampsia | Within one week of delivery
  Hypertension and proteinuria or other organ dysfunction occur after 20 weeks of gestation

SECONDARY OUTCOMES:
Incidence of severe preeclampsia and hypertensive disorders of pregnancy | Within one week of delivery
  Severe preeclampsia or hypertensive disorders of pregnancy occur in pregnant women
Outcome of the fetus | Within one week of delivery
  The incidence of SGA, premature birth and fetal death in utero
Complications of the mother | Within one week of delivery
  The incidence of placental abruption, oligohydramnios, HELLP syndrome, and preeclampsia and postpartum hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Fang He, M.D, Principal Investigator — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Fang He, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No